CLINICAL TRIAL: NCT01558271
Title: A Phase 3 Study of LY2189265 Monotherapy Compared to Placebo and Liraglutide in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2189265 in Japanese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13990; H9X-JE-GBDP (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-03-12; First posted 2012-03-20 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2189265 (Experimental): Once-weekly subcutaneous (SC) injection of 0.75 milligrams (mg) of LY2189265 for 26 weeks of blinded therapy, followed by once-weekly SC injection of 0.75 mg LY2189265 for an additional 26 weeks of open therapy.
  Interventions: Drug: LY2189265
- Placebo/LY2189265 (Placebo Comparator): Once-weekly SC injection of placebo for 26 weeks of blinded therapy, followed by once-weekly SC injection of 0.75 mg LY2189265 for an additional 26 weeks of open therapy.
  Interventions: Drug: LY2189265; Drug: Placebo
- Liraglutide (Active Comparator): Once-daily SC injection of 0.3 mg of Liraglutide for the first week, followed by 0.6 mg of Liraglutide for the second week, and then 0.9 mg of Liraglutide for the remaining 50 weeks of open therapy.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: LY2189265
  Other Names: Dulaglutide
  Arms: LY2189265; Placebo/LY2189265
Drug: Placebo
  Arms: Placebo/LY2189265
Drug: Liraglutide
  Arms: Liraglutide

SUMMARY:
The purpose of this trial is to examine the efficacy and safety of once-weekly LY2189265 in participants with type 2 diabetes mellitus who are not taking oral antidiabetic medication.

DETAILED DESCRIPTION:
Rescue therapy (defined as alternative antihyperglycemic medication use or dose modification of oral antihyperglycemic medication [OAM]) may have been initiated during the planned treatment period if the participant discontinued study drug or met prespecified thresholds for severe, persistent hyperglycemia. Efficacy data, as well as data for hypoglycemic episodes from participants who permanently discontinued study treatment but switched to another diabetes medication and remained in the study, were censored from the point of initiating new treatment onwards.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have had a diagnosis of type 2 diabetes mellitus before screening.
* Participants who have been Oral Antihyperglycemic Medication (OAM)-naïve (diet and exercise only) or been taking OAM monotherapy except for thiazolidinedione (TZD) and are willing to discontinue this medication. Participants taking OAM monotherapy must complete 8-week washout period prior to randomization.
* Participants who are OAM naïve with a screening glycosylated hemoglobin (HbA1c) value of 7.0% to 10.0% and randomization HbA1c value of 7.0% to 10.0%, or who are taking OAM monotherapy with screening HbA1c value of 6.5% to 9.0% and randomization HbA1c value of 7.0% to 10.0%.
* Participants who have a body mass index (BMI) of 18.5 kilograms per meter squared (kg/m^2) to 35.0 kg/m^2.

Exclusion Criteria:

* Participants who have a diagnosis of type 1 diabetes.
* Participants who have previously been treated with any other glucagon-like peptide-1 (GLP-1) analog.
* Participants who have been receiving more than half of the maximum dose of sulfonylureas at screening.
* Participants who have been currently taking insulin or TZD, or have had previous insulin or TZD treatment within 3 months before screening.
* Participants who have obvious clinical signs or symptoms of pancreatitis, a history of chronic pancreatitis or acute pancreatitis at screening, as determined by the investigator. Participants who have a serum amylase concentration ≥3 times the upper limit of the reference range and/or a serum lipase concentration ≥2 times the upper limit of the reference range, as determined by the central laboratory at screening.
* Participants who have self or family history of medullary C-cell hyperplasia, focal hyperplasia, or medullary thyroid carcinoma (MTC).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- Japan (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ishikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yokohama

REFERENCES:
- [Derived] Iwamoto N, Matsui A, Kazama H, Oura T. Subgroup Analysis Stratified by Baseline Pancreatic beta-cell Function in a Japanese Study of Dulaglutide in Patients with Type 2 Diabetes. Diabetes Ther. 2018 Feb;9(1):383-394. doi: 10.1007/s13300-017-0346-4. Epub 2017 Dec 20. PMID 29264713
- [Derived] Suzuki S, Oura T, Takeuchi M, Boye KS. Evaluation of the impact of once weekly dulaglutide on patient-reported outcomes in Japanese patients with type 2 diabetes: comparisons with liraglutide, insulin glargine, and placebo in two randomized studies. Health Qual Life Outcomes. 2017 Jun 12;15(1):123. doi: 10.1186/s12955-017-0696-7. PMID 28606095

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Started | 281 | 70 | 141
Received at Least 1 Dose of Study Drug | 280 | 70 | 137
Completed 26 Weeks | 271 | 63 | 128
Completed | 263 | 59 | 124
Not Completed | 18 | 11 | 17
Not completed — Adverse Event | 6 | 3 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 6 | 12
Not completed — Physician Decision | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study medication.
Groups:
- LY2189265: Once-weekly SC injection of 0.75 mg of LY2189265 for 26 weeks of blinded therapy, followed by once-weekly SC injection of 0.75 mg LY2189265 for an additional 26 weeks of open therapy.
- Total: Total of all reporting groups
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide | Total
Number analyzed (Participants) | 280 | 70 | 137 | 487
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.15 (9.57) | 57.66 (8.34) | 57.91 (10.93) | 57.44 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 15 | 24 | 91
  Male | 228 | 55 | 113 | 396
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 280 | 70 | 137 | 487
Region of Enrollment [Number; unit: participants]
  Japan | 280 | 70 | 137 | 487

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at 26 Weeks
Description: Least squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) analysis with treatment, visit, treatment-by-visit, prestudy therapy (oral antihyperglycemic medication [OAM] yes/no), baseline body mass index (BMI) group (<25 or >=25 kilograms per meter squared [kg/m^2]) as fixed effects, baseline HbA1c as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks
Population: Participants who received at least one dose of study medication with evaluable HbA1c data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- LY2189265: Once-weekly SC injection of 0.75 mg of LY2189265 for 26 weeks of blinded therapy.
- Placebo: Once-weekly SC injection of placebo for 26 weeks of blinded therapy.
- Liraglutide: Once-daily SC injection of 0.3 mg of Liraglutide for the first week, followed by 0.6 mg of Liraglutide for the second week, and then 0.9 mg of Liraglutide for the remaining 24 weeks of open therapy.
Arm/Group | LY2189265 | Placebo | Liraglutide
Number analyzed (Participants) | 280 | 68 | 136
percentage of HbA1c | -1.43 (0.05) | 0.14 (0.10) | -1.33 (0.07)
Statistical Analysis 1: Comparison: LY2189265 vs Placebo; Approximately 490 participants were to be randomized in a 4:1:2 ratio to LY2189265, placebo, or Liraglutide, respectively. This sample size would provide greater than 99% power to demonstrate superiority of LY2189265 to placebo. This computation assumed a true mean difference in HbA1c change from baseline between LY2189265 and placebo being 0.8%, a common standard deviation of 1.1%, a 1-sided significance level of 0.025, and a 9% drop-out rate between randomization and Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.57, 95% CI 2-sided [-1.79 to -1.35]
Statistical Analysis 2: Comparison: LY2189265 vs Liraglutide; Approximately 490 participants were to be randomized in a 4:1:2 ratio to LY2189265, placebo, or Liraglutide, respectively. This sample size would provide >90% power to confirm non-inferiority of LY2189265 to liraglutide by a margin of 0.4%. This computation assumed a true mean difference in HbA1c change from baseline between LY2189265 and Liraglutide being 0%, a common standard deviation of 1.1%, a 1-sided significance level of 0.025, and a 9% drop-out rate between randomization and Week 26; Test type: Non-Inferiority or Equivalence — If the upper limit of the 95% Confidence Interval (CI) was <0.4%, then LY2189265 was declared non-inferior to Liraglutide. If the upper limit of the 95% CI was <0.0%, then LY2189265 was declared superior to liraglutide; p = 0.248, Mixed Models Analysis; LS Mean Difference = -0.10, 95% CI 2-sided [-0.27 to 0.07]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at 52 Weeks
Description: LS means were calculated using MMRM analysis with treatment, visit, treatment-by-visit, prestudy therapy (OAM yes/no), baseline BMI group (<25 or >=25 kg/m^2) as fixed effects, baseline HbA1c as a covariate, and participant as a random effect.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- Liraglutide: Once-daily SC injection of 0.3 mg of Liraglutide for the first week followed by 0.6 mg of Liraglutide for the second week, and then 0.9 mg of Liraglutide for the remaining 50 weeks of open therapy.
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 68 | 136
percentage of HbA1c | -1.39 (0.06) | -1.55 (0.12) | -1.19 (0.08)
Statistical Analysis 1: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.040, Mixed Models Analysis; LS Mean Difference = -0.20, 95% CI 2-sided [-0.39 to -0.01]

3. Secondary Outcome: Percentage of Participants Who Achieved HbA1c <=6.5% or <7%
Description: The percentage of participants achieving HbA1c level less than 7.0% and less than or equal to 6.5% at Week 26 and Week 52 was analyzed with a Cochran-Mantel-Haenszel test stratified by prestudy therapy (OAM yes/no) and baseline BMI group (<25 or >=25 kg/m^2).
Time Frame: Up to 26 and 52 weeks
Population: Participants who were randomized and received at least one dose of study medication with evaluable HbA1c data. Only pre-rescue measurements were used. Missing endpoints were imputed with the last observation carried forward (LOCF), using only postbaseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 68 | 136
percentage of participants
  HbA1c <7%, 26 weeks | 71.4 | 5.9 | 69.1
  HbA1c <=6.5%, 26 weeks | 50.0 | 1.5 | 49.3
  HbA1c <7%, 52 weeks | 67.9 | 70.6 | 60.3
  HbA1c <=6.5%, 52 weeks | 49.3 | 52.9 | 41.2
Statistical Analysis 1: Comparison: LY2189265 vs Placebo/LY2189265; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Treatment comparison for HbA1c <7% at 26 weeks between LY2189265 and placebo; Pairwise comparison was adjusted for prestudy therapy (OAM yes/no), baseline BMI group (<25 / >=25 kg/m^2), and baseline HbA1c group
Statistical Analysis 2: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.608, Cochran-Mantel-Haenszel — Treatment comparison for HbA1c <7% at 26 weeks between LY2189265 and Liraglutide; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: LY2189265 vs Placebo/LY2189265; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Treatment comparison for HbA1c <=6.5% at 26 weeks between LY2189265 and placebo; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.844, Cochran-Mantel-Haenszel — Treatment comparison for HbA1c <=6.5% at 26 weeks between LY2189265 and Liraglutide; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.112, Cochran-Mantel-Haenszel — Treatment comparison for HbA1c <7% at 52 weeks between LY2189265 and Liraglutide; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.103, Cochran-Mantel-Haenszel — Treatment comparison for HbA1c <=6.5% at 52 weeks between LY2189265 and Liraglutide; [statistical method as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) at 26 Weeks and 52 Weeks
Description: LS means were calculated using MMRM analysis with treatment, visit, treatment-by-visit, prestudy therapy (OAM yes/no), baseline BMI group (<25 or >=25 kg/m^2) as fixed effects, baseline FBG as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized and received at least one dose of study medication with evaluable FBG data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 276 | 62 | 134
milligrams per deciliter (mg/dL)
  26 weeks | -39.18 (1.60) | 1.03 (3.30) | -39.75 (2.27)
  52 weeks | -38.93 (1.72) | -40.93 (3.62) | -37.15 (2.47)
Statistical Analysis 1: Comparison: LY2189265 vs Placebo/LY2189265; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison for FBG at 26 weeks between LY2189265 and placebo; LS Mean Difference = -40.21, 95% CI 2-sided [-47.31 to -33.11]
Statistical Analysis 2: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.835, Mixed Models Analysis; Treatment comparison for FBG at 26 weeks between LY2189265 and Liraglutide; LS Mean Difference = 0.57, 95% CI 2-sided [-4.82 to 5.96]
Statistical Analysis 3: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.553, Mixed Models Analysis — Treatment comparison for FBG at 52 weeks between LY2189265 and Liraglutide; LS Mean Difference = -1.77, 95% CI 2-sided [-7.65 to 4.10]

5. Secondary Outcome: Change From Baseline in 7-Point Self-Monitored Blood Glucose (SMBG) at 26 Weeks and 52 Weeks
Description: Participants were to test and record SMBG concentrations in their study diaries before each meal (breakfast, lunch, and dinner), approximately 2 hours after the start of each meal, and at bedtime. LS means were calculated using analysis of covariance (ANCOVA) model with treatment, prestudy therapy (OAM yes/no), and baseline BMI group (<25 or >=25 kg/m^2) as fixed effects and baseline SMBG as a covariate.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who received at least one dose of study medication with evaluable SMBG data. Only pre-rescue measurements were used. Missing endpoints were imputed with the LOCF method, using only postbaseline data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 277 | 69 | 133
milligrams per deciliter (mg/dL)
  Pre-morning meal, 26 weeks | -39.65 (1.55) | -0.15 (3.04) | -34.93 (2.19)
  2 hours post-morning meal, 26 weeks | -69.64 (2.80) | -9.29 (5.48) | -61.67 (3.96)
  Pre-midday meal, 26 weeks | -48.47 (2.05) | 3.91 (4.03) | -45.08 (2.91)
  2 hours post-midday meal, 26 weeks | -67.57 (2.94) | -1.50 (5.77) | -66.71 (4.16)
  Pre-evening meal, 26 weeks | -39.64 (2.15) | 9.25 (4.22) | -36.62 (3.05)
  2 hours post-evening meal | -56.70 (2.83) | 0.93 (5.56) | -53.14 (4.01)
  Bedtime, 26 weeks | -53.39 (2.81) | 4.26 (5.51) | -51.07 (3.94)
  Pre-morning meal, 52 weeks | -37.46 (1.58) | -30.12 (3.10) | -33.41 (2.23)
  2 hours post-morning meal, 52 weeks | -66.96 (2.87) | -65.91 (5.62) | -60.69 (4.06)
  Pre-midday meal, 52 weeks | -47.03 (1.86) | -45.15 (3.64) | -46.25 (2.63)
  2 hours post-midday meal, 52 weeks | -68.21 (2.74) | -58.52 (5.38) | -62.57 (3.88)
  Pre-evening meal, 52 weeks | -41.04 (1.08) | -36.13 (3.70) | -32.86 (2.67)
  2 hours post-evening meal, 52 weeks | -55.01 (2.58) | -55.26 (5.06) | -42.30 (3.65)
  Bedtime, 52 weeks | -55.76 (2.39) | -51.19 (4.69) | -49.10 (3.35)

6. Secondary Outcome: Change From Baseline in Body Weight at 26 Weeks and 52 Weeks
Description: LS means were calculated using MMRM analysis with treatment, visit, treatment-by-visit, prestudy therapy (OAM yes/no), baseline BMI group (<25 or >=25 kg/m^2) as fixed effects, baseline body weight as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who received at least one dose of study medication with evaluable body weight data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 70 | 136
kilograms (kg)
  26 weeks | -0.02 (0.14) | -0.63 (0.29) | -0.36 (0.20)
  52 weeks | -0.17 (0.18) | -1.03 (0.37) | -0.13 (0.26)
Statistical Analysis 1: Comparison: LY2189265 vs Placebo/LY2189265; Test type: Superiority or Other; p = 0.057, Mixed Models Analysis; Treatment comparison for body weight at 26 weeks between LY2189265 and placebo; LS Mean Difference = 0.61, 95% CI 2-sided [-0.02 to 1.23]
Statistical Analysis 2: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.168, Mixed Models Analysis — Treatment comparison for body weight at 26 weeks between LY2189265 and Liraglutide; LS Mean Difference = 0.34, 95% CI 2-sided [-0.14 to 0.82]
Statistical Analysis 3: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.911, Mixed Models Analysis — Treatment comparison for body weight at 52 weeks between LY2189265 and Liraglutide; LS Mean Difference = -0.03, 95% CI 2-sided [-0.64 to 0.57]

7. Secondary Outcome: Change From Baseline in Insulin Sensitivity Using Updated Homeostasis Model Assessment (HOMA 2) at 26 Weeks and 52 Weeks
Description: HOMA 2 quantifies insulin resistance and beta-cell function. HOMA2-S is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin sensitivity (%S) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. Change in insulin sensitivity was assessed based on change from baseline of HOMA2-%S using fasting insulin (FI) and fasting C-peptide (FCP). LS means were calculated using ANCOVA model with treatment, prestudy therapy (OAM yes/no), and baseline BMI group (<25 or >=25 kg/m^2) as fixed effects and baseline HOMA2-%S as a covariate.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized and received at least one dose of study medication with evaluable HOMA2-%S data. Only pre-rescue measurements were used. Missing endpoints were imputed with the LOCF method, using only postbaseline data.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 275 | 62 | 131
percentage of HOMA2
  HOMA2-%S based on FI, 26 weeks (n=254, 57, 115) | -4.83 (2.34) | -2.97 (4.83) | -4.82 (3.43)
  HOMA2-%S based on FCP, 26 weeks (n=275, 62, 131) | -5.48 (1.93) | -6.32 (3.99) | -2.46 (2.75)
  HOMA2-%S based on FI, 52 weeks (n=260, 60, 120) | -7.75 (2.34) | NA (NA) — For ANCOVA analyses at 52 weeks, LS Means were not calculated for the Placebo/LY2189265 group as the purpose of the Week 52 analysis was to evaluate the efficacy and safety of LY2189265 compared with Liraglutide treatment for a full 52 weeks. | -5.26 (3.38)
  HOMA2-%S based on FCP, 52 weeks (n=275, 62, 131) | -11.72 (1.88) | NA (NA) — For ANCOVA analyses at 52 weeks, LS Means were not calculated for the Placebo/LY2189265 group as the purpose of the Week 52 analysis was to evaluate the efficacy and safety of LY2189265 compared with Liraglutide treatment for a full 52 weeks. | -10.68 (2.68)
Statistical Analysis 1: Comparison: LY2189265 vs Placebo/LY2189265; Test type: Superiority or Other; p = 0.723, ANCOVA — Treatment comparison for HOMA2-%S based on fasting insulin at 26 weeks between LY2189265 and placebo; LS Mean Difference = -1.86, 95% CI 2-sided [-12.20 to 8.48]
Statistical Analysis 2: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.998, ANCOVA — Treatment comparison for HOMA2-%S based on fasting insulin at 26 weeks between LY2189265 and Liraglutide; LS Mean Difference = -0.01, 95% CI 2-sided [-7.92 to 7.91]
Statistical Analysis 3: Comparison: LY2189265 vs Placebo/LY2189265; Test type: Superiority or Other; p = 0.848, ANCOVA — Treatment comparison for HOMA2-%S based on fasting C-peptide at 26 weeks between LY2189265 and placebo; LS Mean Difference = 0.83, 95% CI 2-sided [-7.72 to 9.38]
Statistical Analysis 4: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.357, ANCOVA — Treatment comparison for HOMA2-%S based on fasting C-peptide at 26 weeks between LY2189265 and Liraglutide; LS Mean Difference = -3.03, 95% CI 2-sided [-9.48 to 3.42]
Statistical Analysis 5: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.533, ANCOVA — Treatment comparison for HOMA2-%S based on fasting insulin at 52 weeks between LY2189265 and Liraglutide; LS Mean Difference = -2.49, 95% CI 2-sided [-10.35 to 5.36]
Statistical Analysis 6: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.747, ANCOVA — Treatment comparison for HOMA2-%S based on fasting C-peptide at 52 weeks between LY2189265 and Liraglutide; LS Mean Difference = -1.03, 95% CI 2-sided [-7.32 to 5.25]

8. Secondary Outcome: Change From Baseline in Beta-cell Function Using Updated Homeostasis Model Assessment (HOMA 2) at 26 Weeks and 52 Weeks
Description: HOMA 2 quantifies insulin resistance and beta-cell function. HOMA2-B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state beta-cell function (%B) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. Change in beta-cell function was assessed based on change from baseline of HOMA2-%B using fasting insulin (FI) and fasting C-peptide (FCP). LS means were calculated using ANCOVA model with treatment, prestudy therapy (OAM yes/no), and baseline BMI group (<25 or >=25 kg/m^2) as fixed effects and baseline HOMA2-%B as a covariate.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized and received at least one dose of study medication with evaluable HOMA2-%B data. Only pre-rescue measurements were used. Missing endpoints were imputed with the LOCF method, using only postbaseline data.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 275 | 62 | 131
percentage of HOMA2
  HHOMA2-%B based on FI, 26 weeks (n=254, 57, 115) | 28.42 (1.54) | 0.08 (3.14) | 25.35 (2.23)
  HOMA2-%B based on FCP, 26 weeks (n=275, 62, 131) | 27.77 (1.27) | 2.94 (2.61) | 25.86 (1.79)
  HOMA2-%B based on FI, 52 weeks (n=260, 60, 120) | 27.81 (1.39) | NA (NA) — For ANCOVA analyses at 52 weeks, LS Means were not calculated for the Placebo/LY2189265 group as the purpose of the Week 52 analysis was to evaluate the efficacy and safety of LY2189265 compared with Liraglutide treatment for a full 52 weeks. | 25.89 (1.99)
  HOMA2-%B based on FCP, 52 weeks (n=275, 62, 131) | 29.59 (1.37) | NA (NA) — For ANCOVA analyses at 52 weeks, LS Means were not calculated for the Placebo/LY2189265 group as the purpose of the Week 52 analysis was to evaluate the efficacy and safety of LY2189265 compared with Liraglutide treatment for a full 52 weeks. | 28.85 (1.93)
Statistical Analysis 1: Comparison: LY2189265 vs Placebo/LY2189265; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison for HOMA2-%B based on fasting insulin at 26 weeks between LY2189265 and placebo; LS Mean Difference = 28.35, 95% CI 2-sided [21.63 to 35.07]
Statistical Analysis 2: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.242, ANCOVA — Treatment comparison for HOMA2-%B based on fasting insulin at 26 weeks between LY2189265 and Liraglutide; LS Mean Difference = 3.08, 95% CI 2-sided [-2.09 to 8.24]
Statistical Analysis 3: Comparison: LY2189265 vs Placebo/LY2189265; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison for HOMA2-%B based on fasting C-peptide at 26 weeks between LY2189265 and placebo; LS Mean Difference = 24.82, 95% CI 2-sided [19.25 to 30.40]
Statistical Analysis 4: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.376, ANCOVA — Treatment comparison for HOMA2-%B based on fasting C-peptide at 26 weeks between LY2189265 and Liraglutide; LS Mean Difference = 1.91, 95% CI 2-sided [-2.32 to 6.13]
Statistical Analysis 5: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.417, ANCOVA — Treatment comparison for HOMA2-%B based on fasting insulin at 52 weeks between LY2189265 and Liraglutide; LS Mean Difference = 1.91, 95% CI 2-sided [-2.72 to 6.54]
Statistical Analysis 6: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p = 0.753, ANCOVA — Treatment comparison for HOMA2-%B based on fasting C-peptide at 52 weeks between LY2189265 and Liraglutide; LS Mean Difference = 0.73, 95% CI 2-sided [-3.83 to 5.29]

9. Secondary Outcome: Percentage of Participants With Hypoglycemic Episodes
Description: The percentage of participants with hypoglycemic episodes was calculated by dividing the number of participants with at least one hypoglycemic episode over the 26-week or 52-week treatment period by the total number of participants analyzed, multiplied by 100%. All classifications of hypoglycemia (documented symptomatic, asymptomatic, severe, nocturnal, non-nocturnal, probable symptomatic, relative, and unspecified) were included, except for episodes of relative hypoglycemia that were not severe. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks
Population: Participants who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 70 | 137
percentage of participants
  26 weeks | 2.1 | 1.4 | 1.5
  52 weeks | 2.9 | 2.9 | 2.9
Statistical Analysis 1: Comparison: LY2189265 vs Placebo/LY2189265; Test type: Superiority or Other; p > 0.999, Fisher Exact — Treatment comparison at 26 weeks between LY2189265 and placebo
Statistical Analysis 2: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p > 0.999, Fisher Exact — Treatment comparison at 26 weeks between LY2189265 and Liraglutide
Statistical Analysis 3: Comparison: LY2189265 vs Liraglutide; Test type: Superiority or Other; p > 0.999, Fisher Exact — Treatment comparison at 52 weeks between LY2189265 and Liraglutide

10. Secondary Outcome: 30-Day Rate of Hypoglycemic Episodes
Description: The 30-day total hypoglycemia rate over 26 weeks and 52 weeks of treatment is summarized. All classifications of hypoglycemia (documented symptomatic, asymptomatic, severe, nocturnal, non-nocturnal, probable symptomatic, relative, and unspecified) were included, except for episodes of relative hypoglycemia that were not severe. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks
Population: Participants who received at least one dose of study medication. One participant in the Liraglutide reporting group received study drug but discontinued from the study on the same day and, therefore, was not included in the analysis.
Measure: Mean (Standard Deviation); unit: events per participant per 30 days
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 70 | 136
events per participant per 30 days
  26 weeks | 0.01 (0.04) | 0.00 (0.02) | 0.00 (0.02)
  52 weeks | 0.00 (0.02) | 0.01 (0.09) | 0.01 (0.04)

11. Secondary Outcome: Number of Participants With Adjudicated Cardiovascular Events at 26 Weeks and 52 Weeks
Description: Deaths and nonfatal cardiovascular adverse events were adjudicated by a committee of physicians with cardiology expertise external to the Sponsor. The nonfatal cardiovascular events subjected to adjudication included myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions (such as coronary artery bypass graft or percutaneous coronary intervention), and cerebrovascular events including cerebrovascular accident (stroke) and transient ischemic attack. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks
Population: Participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 70 | 137
participants
  26 weeks | 0 | 0 | 0
  52 weeks | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Pulse Rate at 26 Weeks and 52 Weeks
Description: Sitting pulse rate was measured. LS means were calculated using ANCOVA model with treatment, prestudy therapy (OAM yes/no), and baseline BMI group (<25 or >=25 kg/m^2) as fixed effects and baseline pulse rate as a covariate.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized and received at least one dose of study medication with evaluable pulse rate data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 70 | 136
beats per minute (bpm)
  26 weeks | 3.35 (0.45) | 1.49 (0.90) | 4.77 (0.64)
  52 weeks | 3.11 (0.42) | 4.42 (0.86) | 5.13 (0.60)

13. Secondary Outcome: Change From Baseline in Blood Pressure at 26 Weeks and 52 Weeks
Description: Sitting systolic blood pressure (SBP) and sitting diastolic blood pressure (DBP) were measured. LS means were calculated using ANCOVA model with treatment, prestudy therapy (OAM yes/no), and baseline BMI group (<25 or >=25 kg/m^2) as fixed effects and baseline blood pressure as a covariate.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized and received at least one dose of study medication with evaluable blood pressure data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: milliliters of mercury (mmHG)
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 70 | 136
milliliters of mercury (mmHG)
  SBP, 26 weeks | 0.62 (0.62) | 0.53 (1.25) | -2.10 (0.89)
  DBP, 26 weeks | 1.09 (0.39) | 0.29 (0.78) | 0.43 (0.56)
  SBP, 52 weeks | 1.32 (0.66) | 0.37 (1.37) | -1.86 (0.95)
  DBP, 52 weeks | 1.41 (0.41) | 1.16 (0.86) | 1.17 (0.60)

14. Secondary Outcome: Number of Participants With Adjudicated Pancreatitis at 26 Weeks and 52 Weeks
Description: Events of pancreatitis (including suspected pancreatitis and severe or serious abdominal pain) were adjudicated by a committee of expert physicians external to the Sponsor. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks
Population: Participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 70 | 137
participants
  26 weeks | 0 | 0 | 0
  52 weeks | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in Pancreatic Enzymes at 26 Weeks and 52 Weeks
Description: Pancreatic enzyme (lipase and total amylase) concentrations were measured.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized and received at least one dose of study medication with evaluable pancreatic enzyme data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: units/liter
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 275 | 65 | 131
units/liter
  Lipase, 26 weeks | 7.0 [1.0 to 13.0] | 1.0 [-6.0 to 5.0] | 11.0 [5.0 to 21.0]
  Total Amylase, 26 weeks | 7.0 [2.0 to 15.0] | 0.0 [-6.0 to 6.0] | 7.0 [1.0 to 15.0]
  Lipase, 52 weeks | 6.0 [1.0 to 12.0] | 6.0 [2.0 to 12.0] | 9.0 [3.0 to 19.0]
  Total Amylase, 52 weeks | 7.0 [1.0 to 14.0] | 9.0 [3.0 to 14.0] | 6.0 [1.0 to 11.0]

16. Secondary Outcome: Change From Baseline in Serum Calcitonin at 26 Weeks and 52 Weeks
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized and received at least one dose of study medication with evaluable serum calcitonin data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: picograms/milliliter
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 274 | 65 | 131
picograms/milliliter
  26 weeks | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  52 weeks | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

17. Secondary Outcome: Number of Participants With Treatment-Emergent LY2189265 Anti-Drug Antibodies (ADAs) at 26 Weeks and 52 Weeks
Description: A participant was considered to have treatment-emergent LY2189265 ADAs if the participant had at least 1 titer that was treatment-emergent relative to baseline, defined as a 4-fold or greater increase in titer from the baseline measurement.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks
Population: Participants who received at least one dose of study medication and had LY2189265 evaluable ADA data.
Measure: Number; unit: participants
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 279 | 68 | 134
participants
  26 weeks (n=279, 68, 133) | 3 | 0 | 0
  52 weeks (n=279, 68, 134) | 3 | 0 | 0

18. Secondary Outcome: Number of Participants Requiring Additional Intervention Due to Hyperglycemia at 26 Weeks and 52 Weeks
Description: Additional intervention was defined as any additional therapeutic intervention in participants who developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, or initiation of an alternative antihyperglycemic medication following study drug discontinuation. The number of participants requiring additional intervention due to hyperglycemia is summarized cumulatively at 26 and 52 weeks.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks
Population: Participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 280 | 70 | 137
participants
  26 weeks | 0 | 0 | 0
  52 weeks | 0 | 0 | 0

19. Secondary Outcome: Change From Baseline in Electrocardiogram Parameters at 26 Weeks and 52 Weeks
Description: Fridericia Corrected QT (QTcF) Interval and PR Interval are summarized. The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTcF = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. PR is the interval between the P wave and the QRS complex. LS means were calculated using ANCOVA model with treatment as a fixed effect and the baseline ECG parameter as the covariate.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized and received at least one dose of study medication with evaluable ECG data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Number analyzed (Participants) | 274 | 65 | 128
milliseconds (msec)
  QTcF, 26 weeks (n=273, 64, 128) | -2.02 (0.70) | -0.96 (1.44) | -1.89 (1.02)
  QTcF, 52 weeks (n=274, 64, 128) | -2.76 (0.68) | -0.80 (1.41) | -4.35 (1.00)
  PR, 26 weeks (n=269, 65, 126) | 2.20 (0.60) | -0.45 (1.22) | 2.07 (0.88)
  PR, 52 weeks (n=270, 65, 126) | 2.81 (0.82) | 2.60 (1.33) | 3.71 (1.03)

ADVERSE EVENTS:
Arm/Group | LY2189265 | Placebo/LY2189265 | Liraglutide
Serious Adverse Events (participants affected / at risk) | 9/280 | 5/70 | 7/137
Other Adverse Events (participants affected / at risk) | 182/280 | 53/70 | 94/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2189265 (N=280) | Placebo/LY2189265 (N=70) | Liraglutide (N=137)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hiv infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/52 (0) | 1/15 (1) | 0/24 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 (0) | 1/55 (1) | 0/113 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2189265 (N=280) | Placebo/LY2189265 (N=70) | Liraglutide (N=137)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 5 (5) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Eustachian tube obstruction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
Diabetic retinopathy (Eye disorders) | 2 (2) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pingueculitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 9 (10) | 1 (1) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 12 (12) | 0 (0) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 22 (24) | 4 (4) | 11 (11)
Dental caries (Gastrointestinal disorders) | 4 (5) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 20 (23) | 6 (6) | 6 (6)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (3) | 1 (1) | 3 (5)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 17 (25) | 2 (2) | 11 (18)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Radicular cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (6) | 0 (0) | 1 (2)
Application site haematoma (General disorders) | 1 (1) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 3 (3)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site dermatitis (General disorders) | 1 (2) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 4 (5)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 5 (5) | 0 (0) | 5 (6)
Injection site rash (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 3 (3) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (8) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 1 (1)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 5 (5) | 0 (0) | 2 (2)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Anisakiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 7 (9) | 2 (2) | 3 (4)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 7 (7) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 52 (61) | 7 (12) | 24 (34)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Pharyngitis (Infections and infestations) | 3 (3) | 3 (4) | 3 (3)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (3)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 5 (5)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Arteriogram coronary (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 0 (0) | 3 (4)
Blood triglycerides increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 10 (11) | 2 (2) | 3 (3)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pancreatic enzymes increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0/228 (0) | 1/55 (1) | 0/113 (0)
Skin test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 8 (8)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 3 (3) | 6 (7)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/52 (1) | 1/15 (1) | 0/24 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Dizziness exertional (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 5 (5) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (6) | 0 (0) | 2 (3)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/228 (2) | 0/55 (0) | 0/113 (0)
Calculus prostatic (Reproductive system and breast disorders) | 0/228 (0) | 0/55 (0) | 1/113 (1)
Cystocele (Reproductive system and breast disorders) | 0/52 (0) | 1/15 (1) | 0/24 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1/228 (1) | 0/55 (0) | 0/113 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1/52 (1) | 0/15 (0) | 0/24 (0)
Prostatitis (Reproductive system and breast disorders) | 1/228 (1) | 0/55 (0) | 0/113 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0/228 (0) | 0/55 (0) | 1/113 (1)
Rectocele (Reproductive system and breast disorders) | 0/52 (0) | 1/15 (1) | 0/24 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/52 (1) | 0/15 (0) | 0/24 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 0 (0) | 3 (3)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (5)
Denture wearer (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Dental care (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Dental prosthesis placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Intra-cerebral aneurysm operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Large intestinal polypectomy (Surgical and medical procedures) | 3 (3) | 0 (0) | 0 (0)
Limb operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Photocoagulation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Retinal laser coagulation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 2 (3)
Tooth repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 2 (2) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days